CLINICAL TRIAL: NCT02507791
Title: Impact of Fitbit Plus Weight Management Program on Physical Activity and Metabolic Disease in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Farrell, Fellow, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-15-03
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Obesity
Keywords: Fitbit; Obesity; Pediatrics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Fitbit (Experimental): Patients will receive Fitbit in the first phase of the study. In addition to attending weekly weight management classes, patients will wear Fitbit Charge HR devices to track heart rate, "active minutes," steps taken, calories burned, and sleep patterns. Patients will receive weekly phone calls to review this data, and further recommendations will be given to encourage additional physical activity as clinically indicated based on time spent being physically active. The goal will be for individuals to reach 10,000 steps per day, though if subjects are significantly under that goal, realistic goal-setting (recommended increases of physical activity of 10% at a time). Patients will continue this intervention for 12 weeks. After 12 weeks, they will return for reassessment. This coincides with the completion of the weight loss program. Subjects will then be followed remotely for another 12 weeks and phone call interventions will continue before returning for a final study visit.
  Interventions: Other: Fitbit Charge HR plus weekly phone calls to review physical activity data
- Late/Delayed Fitbit (Active Comparator): These subjects will follow a similar pattern except they will not receive Fitbit Charge HR devices until the second phase of the study (specifically after completion of the 12 week weight loss program). In the first phase, these subjects will receive weekly phone calls to offer them the same attention as the experimental group, but instead of reviewing Fitbit data, these subjects will subjectively report their physical activity in minutes and by qualifying their physical activity as light, moderate, or vigorous. These individuals, after 12 weeks, will return for reassessment. At that time, these individuals will receive Fitbits and receive weekly telephone calls for an additional 12 weeks before returning for a final study visit.
  Interventions: Other: Fitbit Charge HR plus weekly phone calls to review physical activity data

INTERVENTIONS:
Other: Fitbit Charge HR plus weekly phone calls to review physical activity data — Patients during weekly Healthy Kids, Healthy Weight classes will also upload their Fitbit data, which will be remotely accessed by the study team and weekly phone calls will be implemented to discuss activity

SUMMARY:
This study is evaluating the feasibility and efficacy of using Fitbit Charge HR devices to remotely track the physical activity of obese pediatric patients who are concurrently enrolled in a comprehensive weight loss intervention program. Patients will receive Fitbit devices and will be called weekly to review their average daily steps and heart rates. Patients will receive the Fitbit either at the beginning of classes or upon completion of classes. Patients will then be followed remotely and called weekly for 12 additional weeks after completing classes. The two groups will be compared to examine for differences.

DETAILED DESCRIPTION:
Patients will be randomly assigned into one of two groups. In the first group, patients will undergo an already established multidisciplinary weight loss intervention program and will also wear Fitbit Charge HR devices. Their data will be regularly uploaded to their Fitbit Dashboard, and this information will be reviewed by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Healthy Kids, Healthy Weight assessment and intervention program
* BMI greater than or equal to the 95th percentile

Exclusion Criteria:

* Compromising medical condition that prevents physical activity (sickle cell disease, severe asthma, fractures, etc)
* Severe intellectual disability
* History of smoking
* Current use of atypical antipsychotics, stimulants

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
BMI z-score | 12 weeks
physical activity as measured by Actigraph | 12 weeks

SECONDARY OUTCOMES:
fasting lipid panel | 12 weeks
fasting glucose | 12 weeks
fasting insulin | 12 weeks
Hemoglobin A1c | 12 weeks
Resting energy expenditure | 12 weeks
  measured using ReeVue indirect calorimeter
Body composition measured by bioelectrial impedance analysis | 12 weeks
Estimation of VO2 max | 12 weeks
  Using recovery heart rate s/p 3 minute step test
Blood pressure | 12 weeks
Average steps taken per day | Daily for 24 weeks
  as measured using Fitbit
Resting heart rate | Daily for 24 weeks
  as measured using Fitbit
Active minutes | Daily for 24 weeks
  as measured using Fitbit
Minutes per day in moderate/vigorous physical heart rate range | Daily for 24 weeks
  as measured using Fitbit
Physical activity self-efficiacy questionnaire | 12 weeks
Responses to sleep questionnaire | 12 weeks
  Assess subjective reports of snoring, restfulness, hours of sleep
Responses to self-image questionnaire (SIQYA) | 12 weeks
  only for individuals greater than 13 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- UH Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States